CLINICAL TRIAL: NCT01784900
Title: Treatment of Gastric Peritoneal Carcinomatosis by Association of Complete Surgical Resection of the Lesions and Intraperitoneal Immunotherapy Using Catumaxomab. A Randomized Phase II Trial.
Brief Title: Treatment of Gastric Peritoneal Carcinomatosis by Association of Complete Surgical Resection of the Lesions and Intraperitoneal Immunotherapy Using Catumaxomab
Acronym: IIPOP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-000475-17; 2011/1793 (Other: CSET number)
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Patients With Gastric Peritoneal Carcinomatosis
MeSH Terms: interventions — catumaxomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Schema B (140µg) (Experimental): * D0 : 20 μg of catumaxomab
  * D2 : 40 μg
  * D4 : 80 μg
  Interventions: Drug: Catumaxomab 140µg
- Schema A (100µg) (Experimental): * D0 : 10 μg of catumaxomab
  * D2 : 30 μg
  * D4 : 60 μg
  Interventions: Drug: Catumaxomab 100µg

INTERVENTIONS:
Drug: Catumaxomab 100µg
  Arms: Schema A (100µg)
Drug: Catumaxomab 140µg
  Arms: Schema B (140µg)

SUMMARY:
Treatment by association of complete surgical excision of the lesions and intraperitoneal immunotherapy using Catumaxomab for patients with gastric peritoneal carcinomatosis

ELIGIBILITY:
Inclusion Criteria:

* consent form signed
* Age >= 18
* Carcinomatosis pre operative known or discivered in intraoperative
* Patients uin good general condition who may have extent surgery associated to specific inflammatory syndrom of immunotherapy
* Patients in good general condition
* Patient insured to social care

Inclusion Criteria (intraoperative):

* Gastric adenocarcinoma with macroscopic peritoneal carcinomatosis (PC) confirmed by extemporaneous histological examination
* CP extension minimal or moderate (peritoneal index ≤ 12).
* Resection of the entire macroscopic lesions detectable (primary tumor, lymph nodes and CP). cleaning D2 lymph node (or D1.5).

Exclusion Criteria:

* Presence of metastasis in reach
* Previous treatment with a non-humanized monoclonal AC- (mice or rat)
* Hypersensitivity to any type of antibody.
* History of cancer within 5 years preceding the entry in the trial other than basal cell skin carcinoma or in situ of the cervix,
* Patients already included in another clinical trial with experimental molecule
* Pregnant, or likely to be or breastfeeding, (Women of childbearing potential should have a pregnancy test (blood) negative 15 days before the date of the surgery) Using of a suitable method of contraception for patients of childbearing age during treatment. adequate contraception Methods includeare: an intrauterine device, hormonal contraception, condom use combined with a spermicide
* Persons deprived of liberty or Trust (including curatorship)
* Unable to undergo medical test for geographical, social or psychological.

Exclusion Criteria (intraoperative):

* Persistent peritoneal lesions visible to the end of the surgery
* Resection of the tail of the pancreas or pancreatic break (because no drainage post-op); break pleural (for K cardia)
* Presence of metastasis in reach during surgery (except for ovarian metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | every 3 months for the first two years

SECONDARY OUTCOMES:
Progression Free Survival | every 3 months for the first two years then every 4 months on year 3 then every 6 months on year 4 and 5

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, Val de Marne, France